CLINICAL TRIAL: NCT06991673
Title: Adolescent Surgery Roadmap Feasibility and Acceptability Study
Acronym: Ane-Roadmap
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sydney Brown, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00265431
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Surgical Procedures
Keywords: positive psychology; mobile health; surgical recovery; adolescent; caregiver; pediatric surgery; mobile health intervention; positive psychology intervention
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician will be masked. The research assistant performing the chart review of the electronic health record will be masked. The PI will be masked, except during the qualitative interviews in which masking would be impossible. Care provider will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive Activity Interventions + Surveys (Active Comparator): Intervention arm participants will complete one of eight positive activities within the Ane-Roadmap App either as individuals or as an adolescent-caregiver team. Positive activities include gratitude journaling, planning positive experiences, savoring, identifying personal strengths, performing acts of kindness, love letters, engaging with beauty, and positive piggy bank. Participants in the intervention group will receive reminders to complete activities as an individual and as an adolescent-caregiver team. Participants will denote with a checkbox whether intervention activities were completed as an individual vs. as an adolescent-caregiver team.
  Participants in the control arm will have access to the Ane-Roadmap app, however all intervention activities will be turned off.
  Both control and intervention groups will complete daily and weekly surveys via links embedded within the Roadmap app. Reminders will be sent to participants to complete surveys each day.
  Interventions: Behavioral: Behavioral Treatment
- Surveys Only (No Intervention): Control arm participants will not have access to the positive psychology interventions activities within the Ane-Roadmap app. They will only complete daily and weekly surveys.

INTERVENTIONS:
Behavioral: Behavioral Treatment — Positive Activity Interventions within Ane-Roadmap App
  Positive Piggy Bank - Capture happy moments by mentally savoring them, recording details, and depositing them into a "piggy bank". Open it when you need a boost.
  Gratitude Diary - Write two unique things daily for which you're grateful. Smile as you record them to enhance gratitude.
  Savoring - Each day, spend 2-3 minutes fully enjoying two positive experiences. Log them for reflection.
  Pleasant Activity Scheduling - Plan and engage in enjoyable activities at least twice weekly. Treat them as important appointments.
  Random Acts of Kindness - Perform five intentional kind acts in a day, four for others and one for yourself.
  Signature Strengths - Use a personal strength in a new way daily and reflect on its impact.
  Love Letter - Express deep appreciation to a loved one in a heartfelt letter and share it with them.
  Engaging with Beauty - Keep a log of beautiful moments in nature, art, or human kindness.
  Other Names: Positive Activity Exercises
  Arms: Positive Activity Interventions + Surveys

SUMMARY:
The goal of this clinical trial is to test the feasibility and acceptability of using a mobile health app, Ane-Roadmap, designed to support adolescents (ages 12-17) undergoing painful surgeries and their caregivers. The main questions it aims to answer are:

* Can adolescent surgery patients and their caregivers be successfully enrolled in the study, with at least 40% of those invited choosing to participate?
* Will participants actively use the mobile app, completing at least two activities per week for at least half of the study period, either individually and/or as a caregiver-adolescent pair?

Participants will:

* Use the Ane-Roadmap app during their post-surgery recovery period to complete resilience-building activities aimed at improving wellbeing
* Use the app either individually or together as a caregiver-adolescent pair.
* Complete surveys regarding risk factors for adverse postsurgical pain outcomes and physical and psychological symptoms experienced postoperatively
* Some participants will complete a semi-structured interview in which experiences with the study and intervention activities will be elicited

ELIGIBILITY:
Inclusion Criteria (Adolescent Patient):

* Patient is aged 12-17 years on the date of surgery
* Surgery is a scheduled surgery (non-emergency)
* Surgery is occurring within the University of Michigan hospital system (University Hospital, C.S. Mott Children's Hospital, Brighton Ambulatory Surgery Center, East Ann Arbor Ambulatory Surgery Center)
* Participants are able to enroll within 1-2 weeks of surgery
* Patient and caregiver must be willing to participate
* Adolescent and caregiver must have a compatible smartphone and/or tablet with internet access and be willing to download an app
* Eligible patient is able to sign/assent form
* Adolescent-caregiver dyad has at least one risk factor for adverse post-operative pain outcomes based on pre-enrollment screening (e.g., worries about managing pain, return to normal activities, limitations in doing desired activities, trouble with sleep)

Inclusion Criteria (Caregiver):

* Patient and caregiver must be willing to participate
* Caregiver must be providing at least 50% of the patient's postsurgical caregiving
* Caregivers agree to provide informed consent that is in regulatory compliance and IRBMED-approved and also in accordance with institutional guidelines
* Adolescent and caregiver must have a compatible smartphone and/or tablet with internet access and be willing to download an app

Exclusion Criteria (Adolescent Patient):

* Adolescent or caregiver are unable to complete intervention activities or surveys in spoken or written English
* Significant developmental delay, making it impossible for the participant to use an app to complete interventions or answer survey questions
* Foster children or wards of the state are not eligible for inclusion
* Hardware removal or debridement surgery (not considered as painful as other orthopedic surgeries)
* Scoliosis surgery (due to extended longitudinal relationship with surgeon)
* Concurrent participation in another behavioral/self-management intervention trial
* Any impairment, activity, or situation that in the judgment of the Study Coordinator or Principal would make it inappropriate for the subject to participate

Exclusion Criteria (Caregiver):

* Significant developmental delay, making it impossible for the participant to use an app to complete interventions or answer survey questions
* Adolescent or caregiver are unable to complete intervention activities or surveys in spoken or written English
* Any impairment, activity, or situation that in the judgment of the Study Coordinator or Principal would make it inappropriate for the subject to participate

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Potential (Feasibility) | Up to 74 days (60 days post-surgery)
  The percent of eligible dyads willing to enroll (N subjects enrolled / N subjects successfully reached). This information will be derived from recruitment data. The threshold for success is that 40% of eligible dyads enroll.
Module Engagement (Feasibility) | Up to 74 days (60 days post-surgery)
  The number of days each week a Roadmap intervention module is used each week. This will be derived from app usage data. Threshold for success: Completion of any intervention module at least twice weekly for 70% of the study weeks as an individual or adolescent-caregiver team.
Module Engagement (Feasibility) | Up to 74 days (60 days post-surgery)
  The number of days each week a Roadmap intervention module is used as an adolescent-caregiver team each week. This will be derived from app usage data. Threshold for success: 2) 50% of participants will complete Roadmap intervention activities as a team at least one time for 50% of the study weeks.

SECONDARY OUTCOMES:
Adolescent Global Health | Up to 74 days (60 days post-surgery)
  Adolescent Global Health, assessed by Patient-Reported Outcomes Measurement Information System Pediatric Profile-25 (Minimum value: 12, Maximum value: 120). Higher scores on positive domains (Physical Function and Peer Relationships) = Better outcome. Higher scores on negative domains (Anxiety, Depressive Symptoms, Fatigue, Pain Interference, Pain Intensity) = Worse outcome.
Caregiver Global Health | Up to 74 days (60 days post-surgery)
  Caregiver Global Health assessed using Patient-Reported Outcomes Measurement Information System 29+2 Profile Version 2.1 (Minimum score: 16, Maximum score 160). Higher scores on positive domains (Physical Function, Ability to Participate in Social Roles and Activities) = Better outcome. Higher scores on negative domains (Anxiety, Depression, Fatigue, Pain Interference, Sleep Disturbance, Pain Intensity) = Worse outcome.
Adolescent pain intensity | Up to 74 days (60 days post-surgery)
  Adolescent pain intensity, assessed using Patient-Reported Outcomes Measurement Information System Pediatric Pain Intensity (Minimum value: 0, Maximum value: 10). Higher scores indicate a worse outcome, representing greater pain intensity.
Adolescent Pain Interference | Up to 74 days (60 days post-surgery)
  Adolescent pain interference, assessed using Patient-Reported Outcomes Measurement Information System Pediatric Pain Interference Short Form 8a (Minimum value: 0, Maximum value: 10). Higher scores indicate a worse outcome, representing greater interference of pain with daily activities and functioning.
Adolescent Mood | Up to 74 days (60 days post-surgery)
  Adolescent mood, assessed using Patient-Reported Outcomes Measurement Information System Pediatric Depressive Symptoms - Mood Subscale (minimum value: 4, Maximum value: 20). Higher scores indicate a worse outcome, representing greater depressive symptoms.
Adolescent anxiety | Up to 74 days (60 days post-surgery)
  Adolescent anxiety, assessed using Patient-Reported Outcomes Measurement Information System Pediatric Anxiety - Anxiety Subscale (Minimum value: 4, Maximum value: 20). Higher scores indicate a worse outcome, reflecting greater anxiety symptoms.
Caregiver anxiety | Up to 74 days (60 days post-surgery)
  Caregiver anxiety, assessed using Patient-Reported Outcomes Measurement Information System Anxiety Subscale (Minimum value: 4, Maximum value: 20). Higher scores indicate a worse outcome, reflecting greater anxiety symptoms.
Caregiver mood | Up to 74 days (60 days post-surgery)
  Caregiver mood, assessed using Patient-Reported Outcomes Measurement Information System Mood Subscale (Minimum value: 4, Maximum value: 20). Higher scores indicate a worse outcome, reflecting greater negative mood symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Brown, MD PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Michigan Medicine- East Ann Arbor Ambulatory Surgery and Medical Procedures Center, Ann Arbor, Michigan
  - University of Michigan affiliated hospitals, Ann Arbor, Michigan
  - Michigan Medicine- Brighton Center for Specialty Care, Brighton, Michigan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary results have been published in a peer-reviewed journal. Study data that is stored at the University of Michigan will be available to the research community in perpetuity.
Access Criteria: All deidentified study data that are not designated as restricted use will be made available on request by contacting the PI or The University of Michigan Department of Anesthesiology. Users must complete a mutually agreed upon data sharing plan, be qualified and approved by the University of Michigan, and agree to the Terms of Use. These processes are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.

REFERENCES:
- [Background] Whittle R, Mansell G, Jellema P, van der Windt D. Applying causal mediation methods to clinical trial data: What can we learn about why our interventions (don't) work? Eur J Pain. 2017 Apr;21(4):614-622. doi: 10.1002/ejp.964. Epub 2016 Oct 14. PMID 27739626
- [Background] Valeri L, Vanderweele TJ. Mediation analysis allowing for exposure-mediator interactions and causal interpretation: theoretical assumptions and implementation with SAS and SPSS macros. Psychol Methods. 2013 Jun;18(2):137-50. doi: 10.1037/a0031034. Epub 2013 Feb 4. PMID 23379553
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Bryant FB. A four-factor model of perceived control: Avoiding, coping, obtaining, and savoring. J Pers. 1989;57(4):773-797.
- [Background] Kashdan TB, Uswatte G, Julian T. Gratitude and hedonic and eudaimonic well-being in Vietnam war veterans. Behav Res Ther. 2006 Feb;44(2):177-99. doi: 10.1016/j.brat.2005.01.005. PMID 16389060
- [Background] Emmons RA, McCullough ME. Counting blessings versus burdens: an experimental investigation of gratitude and subjective well-being in daily life. J Pers Soc Psychol. 2003 Feb;84(2):377-89. doi: 10.1037//0022-3514.84.2.377. PMID 12585811
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Pennarola BW, Rodday AM, Mayer DK, Ratichek SJ, Davies SM, Syrjala KL, Patel S, Bingen K, Kupst MJ, Schwartz L, Guinan EC, Hibbard JH, Parsons SK; HSCT-CHESS Study. Factors associated with parental activation in pediatric hematopoietic stem cell transplant. Med Care Res Rev. 2012 Apr;69(2):194-214. doi: 10.1177/1077558711431460. Epub 2011 Dec 26. PMID 22203645
- [Background] Fauer A, Hoodin F, Byrd M, et al. The role of family caregiving in adult and pediatric allogeneic hematopoietic cell transplantation: Using health information technology to advance patient-centered care. Biol Blood Marrow Transplant. 2018;24(3):S484-S485.
- [Background] Runaas L, Hoodin F, Kentor R, et al. User-centered design and development of a personalized mobile health application for adult HCT patients in the inpatient setting. Biol Blood Marrow Transplant. 2017;23(3):S419-S420.
- [Background] Runaas L, Hoodin F, Munaco A, Fauer A, Sankaran R, Churay T, Mohammed S, Seyedsalehi S, Chappell G, Carlozzi N, Fetters MD, Kentor R, McDiarmid L, Brookshire K, Warfield C, Byrd M, Kaziunas S, Maher M, Magenau J, An L, Cohn A, Hanauer DA, Choi SW. Novel Health Information Technology Tool Use by Adult Patients Undergoing Allogeneic Hematopoietic Cell Transplantation: Longitudinal Quantitative and Qualitative Patient-Reported Outcomes. JCO Clin Cancer Inform. 2018 Dec;2:1-12. doi: 10.1200/CCI.17.00110. PMID 30652535
- [Background] Runaas L, Hanauer D, Maher M, Bischoff E, Fauer A, Hoang T, Munaco A, Sankaran R, Gupta R, Seyedsalehi S, Cohn A, An L, Tewari M, Choi SW. BMT Roadmap: A User-Centered Design Health Information Technology Tool to Promote Patient-Centered Care in Pediatric Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2017 May;23(5):813-819. doi: 10.1016/j.bbmt.2017.01.080. Epub 2017 Jan 27. PMID 28132870
- [Background] Runaas L, Bischoff E, Hoodin F, et al. A novel health informatics tool to improve caregiver activation: Findings from pediatric BMT in a hospital-based setting. Blood. 2016;128(22):2382-2382.
- [Background] Grossman LV, Choi SW, Collins S, Dykes PC, O'Leary KJ, Rizer M, Strong P, Yen PY, Vawdrey DK. Implementation of acute care patient portals: recommendations on utility and use from six early adopters. J Am Med Inform Assoc. 2018 Apr 1;25(4):370-379. doi: 10.1093/jamia/ocx074. PMID 29040634
- [Background] Kaziunas E, Hanauer DA, Ackerman MS, Choi SW. Identifying unmet informational needs in the inpatient setting to increase patient and caregiver engagement in the context of pediatric hematopoietic stem cell transplantation. J Am Med Inform Assoc. 2016 Jan;23(1):94-104. doi: 10.1093/jamia/ocv116. Epub 2015 Oct 28. PMID 26510878
- [Background] Maher M, Kaziunas E, Ackerman M, Derry H, Forringer R, Miller K, O'Reilly D, An LC, Tewari M, Hanauer DA, Choi SW. User-Centered Design Groups to Engage Patients and Caregivers with a Personalized Health Information Technology Tool. Biol Blood Marrow Transplant. 2016 Feb;22(2):349-358. doi: 10.1016/j.bbmt.2015.08.032. Epub 2015 Sep 5. PMID 26343948
- [Background] Choi SW, Chang L, Hanauer DA, Shaffer-Hartman J, Teitelbaum D, Lewis I, Blackwood A, Akcasu N, Steel J, Christensen J, Niedner MF. Rapid reduction of central line infections in hospitalized pediatric oncology patients through simple quality improvement methods. Pediatr Blood Cancer. 2013 Feb;60(2):262-9. doi: 10.1002/pbc.24187. Epub 2012 Apr 22. PMID 22522576
- [Background] Büyüktür AG, Ackerman MS. Issues and opportunities in transitions from speciality care: a field study of bone marrow transplant. Behav Inf Technol. 2015;34(6):566-584.
- [Background] Kubiak RM, Dinh D, Carlozzi NE, Clauw D, Waljee JF, Brown SE. Feasibility and Acceptability of Mobile Technologies for Post-Operative Data Collection in Adolescents and Caregivers. Presented at: Society for Pediatric Anesthesiology; March 2024; Anaheim, CA.
- [Background] Hassett AL, Finan PH. The Role of Resilience in the Clinical Management of Chronic Pain. Curr Pain Headache Rep. 2016 Jun;20(6):39. doi: 10.1007/s11916-016-0567-7. PMID 27115770
- [Background] Bolier L, Haverman M, Westerhof GJ, Riper H, Smit F, Bohlmeijer E. Positive psychology interventions: a meta-analysis of randomized controlled studies. BMC Public Health. 2013 Feb 8;13:119. doi: 10.1186/1471-2458-13-119. PMID 23390882
- [Background] Sin NL, Lyubomirsky S. Enhancing well-being and alleviating depressive symptoms with positive psychology interventions: a practice-friendly meta-analysis. J Clin Psychol. 2009 May;65(5):467-87. doi: 10.1002/jclp.20593. PMID 19301241
- [Background] Porter LS, Keefe FJ, Garst J, McBride CM, Baucom D. Self-efficacy for managing pain, symptoms, and function in patients with lung cancer and their informal caregivers: associations with symptoms and distress. Pain. 2008 Jul 15;137(2):306-315. doi: 10.1016/j.pain.2007.09.010. Epub 2007 Oct 17. PMID 17942229
- [Background] Keefe FJ, Ahles TA, Porter LS, Sutton LM, McBride CM, Pope MS, McKinstry ET, Furstenberg CP, Dalton J, Baucom DH. The self-efficacy of family caregivers for helping cancer patients manage pain at end-of-life. Pain. 2003 May;103(1-2):157-62. doi: 10.1016/s0304-3959(02)00448-7. PMID 12749970
- [Background] Northouse LL, Katapodi MC, Schafenacker AM, Weiss D. The impact of caregiving on the psychological well-being of family caregivers and cancer patients. Semin Oncol Nurs. 2012 Nov;28(4):236-45. doi: 10.1016/j.soncn.2012.09.006. PMID 23107181
- [Background] Badr H, Yeung C, Lewis MA, Milbury K, Redd WH. An observational study of social control, mood, and self-efficacy in couples during treatment for head and neck cancer. Psychol Health. 2015;30(7):783-802. doi: 10.1080/08870446.2014.994633. Epub 2015 Jan 2. PMID 25471820
- [Background] Jackson SE, Steptoe A, Wardle J. The influence of partner's behavior on health behavior change: the English Longitudinal Study of Ageing. JAMA Intern Med. 2015 Mar;175(3):385-92. doi: 10.1001/jamainternmed.2014.7554. PMID 25599511
- [Background] Logan DE, Scharff L. Relationships between family and parent characteristics and functional abilities in children with recurrent pain syndromes: an investigation of moderating effects on the pathway from pain to disability. J Pediatr Psychol. 2005 Dec;30(8):698-707. doi: 10.1093/jpepsy/jsj060. Epub 2005 Aug 10. PMID 16093517
- [Background] Chambers CT. The Role of Family Factors in Pediatric Pain. In: Pediatric Pain: Biological and Social Context. (McGrath PJ FGA, ed.). IASP Press; 2003:99-130.
- [Background] Palermo TM, Valrie CR, Karlson CW. Family and parent influences on pediatric chronic pain: a developmental perspective. Am Psychol. 2014 Feb-Mar;69(2):142-52. doi: 10.1037/a0035216. PMID 24547800
- [Background] Palermo TM, Holley AL. The importance of the family environment in pediatric chronic pain. JAMA Pediatr. 2013 Jan;167(1):93-4. doi: 10.1001/jamapediatrics.2013.428. No abstract available. PMID 23403868
- [Background] Hoftun GB, Romundstad PR, Rygg M. Association of parental chronic pain with chronic pain in the adolescent and young adult: family linkage data from the HUNT Study. JAMA Pediatr. 2013 Jan;167(1):61-9. doi: 10.1001/jamapediatrics.2013.422. PMID 23403843
- [Background] Palermo TM, Chambers CT. Parent and family factors in pediatric chronic pain and disability: an integrative approach. Pain. 2005 Dec 15;119(1-3):1-4. doi: 10.1016/j.pain.2005.10.027. Epub 2005 Nov 18. No abstract available. PMID 16298492
- [Background] Alderfer MA, Fiese BH, Gold JI, Cutuli JJ, Holmbeck GN, Goldbeck L, Chambers CT, Abad M, Spetter D, Patterson J. Evidence-based assessment in pediatric psychology: family measures. J Pediatr Psychol. 2008 Oct;33(9):1046-61; discussion 1062-4. doi: 10.1093/jpepsy/jsm083. Epub 2007 Sep 28. PMID 17905801
- [Background] Lewandowski AS, Palermo TM, Stinson J, Handley S, Chambers CT. Systematic review of family functioning in families of children and adolescents with chronic pain. J Pain. 2010 Nov;11(11):1027-38. doi: 10.1016/j.jpain.2010.04.005. PMID 21055709
- [Background] Garlo K, O'Leary JR, Van Ness PH, Fried TR. Burden in caregivers of older adults with advanced illness. J Am Geriatr Soc. 2010 Dec;58(12):2315-22. doi: 10.1111/j.1532-5415.2010.03177.x. Epub 2010 Nov 18. PMID 21087225
- [Background] Fried TR, Bradley EH, O'Leary JR, Byers AL. Unmet desire for caregiver-patient communication and increased caregiver burden. J Am Geriatr Soc. 2005 Jan;53(1):59-65. doi: 10.1111/j.1532-5415.2005.53011.x. PMID 15667377
- [Background] Coyne JC, Rohrbaugh MJ, Shoham V, Sonnega JS, Nicklas JM, Cranford JA. Prognostic importance of marital quality for survival of congestive heart failure. Am J Cardiol. 2001 Sep 1;88(5):526-9. doi: 10.1016/s0002-9149(01)01731-3. PMID 11524062
- [Background] Antonucci TC, Birditt KS, Webster NJ. Social relations and mortality: a more nuanced approach. J Health Psychol. 2010 Jul;15(5):649-59. doi: 10.1177/1359105310368189. PMID 20603288
- [Background] Birditt K, Antonucci TC. Life sustaining irritations? Relationship quality and mortality in the context of chronic illness. Soc Sci Med. 2008 Oct;67(8):1291-9. doi: 10.1016/j.socscimed.2008.06.029. Epub 2008 Jul 26. PMID 18662845
- [Background] Cohen S. Psychosocial models of the role of social support in the etiology of physical disease. Health Psychol. 1988;7(3):269-97. doi: 10.1037//0278-6133.7.3.269. PMID 3289916
- [Background] Hooker SA, Grigsby ME, Riegel B, Bekelman DB. The Impact of Relationship Quality on Health-Related Outcomes in Heart Failure Patients and Informal Family Caregivers: An Integrative Review. J Cardiovasc Nurs. 2015 Jul-Aug;30(4 Suppl 1):S52-63. doi: 10.1097/JCN.0000000000000270. PMID 25955196
- [Background] Fauth E, Hess K, Piercy K, Norton M, Corcoran C, Rabins P, Lyketsos C, Tschanz J. Caregivers' relationship closeness with the person with dementia predicts both positive and negative outcomes for caregivers' physical health and psychological well-being. Aging Ment Health. 2012;16(6):699-711. doi: 10.1080/13607863.2012.678482. PMID 22548375
- [Background] Williamson GM, Schulz R. Relationship orientation, quality of prior relationship, and distress among caregivers of Alzheimer's patients. Psychol Aging. 1990 Dec;5(4):502-9. doi: 10.1037//0882-7974.5.4.502. PMID 2278672
- [Background] Kramer BJ. Marital history and the prior relationship as predictors of positive and negative outcomes among wife caregivers. Fam Relat. 1993;42(4):367.
- [Background] Walker AJ, Shin HY, Bird DN. Perceptions of relationship change and caregiver satisfaction. Fam Relat. 1990;39(2):147.
- [Background] Perren S, Schmid R, Herrmann S, Wettstein A. The impact of attachment on dementia-related problem behavior and spousal caregivers' well-being. Attach Hum Dev. 2007 Jun;9(2):163-78. doi: 10.1080/14616730701349630. PMID 17508315
- [Background] Norton MC, Piercy KW, Rabins PV, Green RC, Breitner JC, Ostbye T, Corcoran C, Welsh-Bohmer KA, Lyketsos CG, Tschanz JT. Caregiver-recipient closeness and symptom progression in Alzheimer disease. The Cache County Dementia Progression Study. J Gerontol B Psychol Sci Soc Sci. 2009 Sep;64(5):560-8. doi: 10.1093/geronb/gbp052. Epub 2009 Jun 29. PMID 19564210
- [Background] Whitlatch CJ, Schur D, Noelker LS, Ejaz FK, Looman WJ. The stress process of family caregiving in institutional settings. Gerontologist. 2001 Aug;41(4):462-73. doi: 10.1093/geront/41.4.462. PMID 11490044
- [Background] Burgener S, Twigg P. Relationships among caregiver factors and quality of life in care recipients with irreversible dementia. Alzheimer Dis Assoc Disord. 2002 Apr-Jun;16(2):88-102. doi: 10.1097/00002093-200204000-00006. PMID 12040304
- [Background] Rozwadowski M, Dittakavi M, Mazzoli A, Hassett AL, Braun T, Barton DL, Carlozzi N, Sen S, Tewari M, Hanauer DA, Choi SW. Promoting Health and Well-Being Through Mobile Health Technology (Roadmap 2.0) in Family Caregivers and Patients Undergoing Hematopoietic Stem Cell Transplantation: Protocol for the Development of a Mobile Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 18;9(9):e19288. doi: 10.2196/19288. PMID 32945777
- [Background] Griffin JM, Meis LA, MacDonald R, Greer N, Jensen A, Rutks I, Wilt TJ. Effectiveness of family and caregiver interventions on patient outcomes in adults with cancer: a systematic review. J Gen Intern Med. 2014 Sep;29(9):1274-82. doi: 10.1007/s11606-014-2873-2. Epub 2014 May 20. PMID 24841557
- [Background] Juth V, Silver RC, Sender L. The shared experience of adolescent and young adult cancer patients and their caregivers. Psychooncology. 2015 Dec;24(12):1746-53. doi: 10.1002/pon.3785. Epub 2015 Mar 25. PMID 25808790
- [Background] Stefanut AM, Vintila M, Tudorel OI. The Relationship of Dyadic Coping With Emotional Functioning and Quality of the Relationship in Couples Facing Cancer-A Meta-Analysis. Front Psychol. 2021 Jan 8;11:594015. doi: 10.3389/fpsyg.2020.594015. eCollection 2020. PMID 33488460
- [Background] Rusu PP, Bodenmann G, Kayser K. Cognitive emotion regulation and positive dyadic outcomes in married couples. J Soc Pers Relat. 2019;36(1):359-376.
- [Background] Bakker D, Kazantzis N, Rickwood D, Rickard N. Mental Health Smartphone Apps: Review and Evidence-Based Recommendations for Future Developments. JMIR Ment Health. 2016 Mar 1;3(1):e7. doi: 10.2196/mental.4984. PMID 26932350
- [Background] Gupta V, Raj M, Hoodin F, Yahng L, Braun T, Choi SW. Electronic Health Record Portal Use by Family Caregivers of Patients Undergoing Hematopoietic Cell Transplantation: United States National Survey Study. JMIR Cancer. 2021 Mar 9;7(1):e26509. doi: 10.2196/26509. PMID 33687332
- [Background] Shin JY, Chaar D, Davis C, Choi SW, Lee HR. Every cloud has a silver lining: Exploring experiential knowledge and assets of family caregivers. Proc ACM Hum Comput Interact. 2021;5(CSCW2):1-25.
- [Background] Shin JY, Choi SW. Online interventions geared toward increasing resilience and reducing distress in family caregivers. Curr Opin Support Palliat Care. 2020 Mar;14(1):60-66. doi: 10.1097/SPC.0000000000000481. PMID 31842019
- [Background] Shin JY, Chaar D, Kedroske J, Vue R, Chappell G, Mazzoli A, Hassett AL, Hanauer DA, Park SY, Debra B, Choi SW. Harnessing mobile health technology to support long-term chronic illness management: exploring family caregiver support needs in the outpatient setting. JAMIA Open. 2020 Dec 5;3(4):593-601. doi: 10.1093/jamiaopen/ooaa053. eCollection 2020 Dec. PMID 33758797
- [Background] Shin JY, Kang TI, Noll RB, Choi SW. Supporting Caregivers of Patients With Cancer: A Summary of Technology-Mediated Interventions and Future Directions. Am Soc Clin Oncol Educ Book. 2018 May 23;38:838-849. doi: 10.1200/EDBK_201397. PMID 30231412
- [Background] Shin JY, Kedroske J, Vue R, et al. Design considerations for family-centered health management. In: Proceedings of the 17th ACM Conference on Interaction Design and Children. ACM; 2018. doi:10.1145/3202185.3210781
- [Background] Maher M, Hanauer DA, Kaziunas E, Ackerman MS, Derry H, Forringer R, Miller K, O'Reilly D, An L, Tewari M, Choi SW. A Novel Health Information Technology Communication System to Increase Caregiver Activation in the Context of Hospital-Based Pediatric Hematopoietic Cell Transplantation: A Pilot Study. JMIR Res Protoc. 2015 Oct 27;4(4):e119. doi: 10.2196/resprot.4918. PMID 26508379
- [Background] Kedroske J, Koblick S, Chaar D, Mazzoli A, O'Brien M, Yahng L, Vue R, Chappell G, Shin JY, Hanauer DA, Choi SW. Development of a National Caregiver Health Survey for Hematopoietic Stem Cell Transplant: Qualitative Study of Cognitive Interviews and Verbal Probing. JMIR Form Res. 2020 Jan 23;4(1):e17077. doi: 10.2196/17077. PMID 32012037
- [Background] Johnson CM, Johnson TR, Zhang J. A user-centered framework for redesigning health care interfaces. J Biomed Inform. 2005 Feb;38(1):75-87. doi: 10.1016/j.jbi.2004.11.005. PMID 15694887
- [Background] Chaar D, Shin JY, Mazzoli A, Vue R, Kedroske J, Chappell G, Hanauer DA, Barton D, Hassett AL, Choi SW. A Mobile Health App (Roadmap 2.0) for Patients Undergoing Hematopoietic Stem Cell Transplant: Qualitative Study on Family Caregivers' Perspectives and Design Considerations. JMIR Mhealth Uhealth. 2019 Oct 24;7(10):e15775. doi: 10.2196/15775. PMID 31651402
- [Background] Gilley KN, Baroudi L, Yu M, Gainsburg I, Reddy N, Bradley C, Cislo C, Rozwadowski ML, Clingan CA, DeMoss MS, Churay T, Birditt K, Colabianchi N, Chowdhury M, Forger D, Gagnier J, Zernicke RF, Cunningham JL, Cain SM, Tewari M, Choi SW. Risk Factors for COVID-19 in College Students Identified by Physical, Mental, and Social Health Reported During the Fall 2020 Semester: Observational Study Using the Roadmap App and Fitbit Wearable Sensors. JMIR Ment Health. 2022 Feb 10;9(2):e34645. doi: 10.2196/34645. PMID 34992051
- [Background] Fauer AJ, Hoodin F, Lalonde L, Errickson J, Runaas L, Churay T, Seyedsalehi S, Warfield C, Chappell G, Brookshire K, Chaar D, Shin JY, Byrd M, Magenau J, Hanauer DA, Choi SW. Impact of a health information technology tool addressing information needs of caregivers of adult and pediatric hematopoietic stem cell transplantation patients. Support Care Cancer. 2019 Jun;27(6):2103-2112. doi: 10.1007/s00520-018-4450-4. Epub 2018 Sep 20. PMID 30232587
- [Background] Carlozzi NE, Kallen MA, Sander AM, Brickell TA, Lange RT, French LM, Ianni PA, Miner JA, Hanks R. The Development of a New Computer Adaptive Test to Evaluate Anxiety in Caregivers of Individuals With Traumatic Brain Injury: TBI-CareQOL Caregiver-Specific Anxiety. Arch Phys Med Rehabil. 2019 Apr;100(4S):S22-S30. doi: 10.1016/j.apmr.2018.05.027. Epub 2018 Jun 26. PMID 29958902
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Tugade MM, Fredrickson BL, Barrett LF. Psychological resilience and positive emotional granularity: examining the benefits of positive emotions on coping and health. J Pers. 2004 Dec;72(6):1161-90. doi: 10.1111/j.1467-6494.2004.00294.x. PMID 15509280
- [Background] Smeallie E, Rosenthal L, Johnson A, Roslin C, Hassett AL, Choi SW. Enhancing Resilience in Family Caregivers Using an mHealth App. Appl Clin Inform. 2022 Oct;13(5):1194-1206. doi: 10.1055/a-1967-8721. Epub 2022 Oct 25. PMID 36283418
- [Background] Joyce S, Shand F, Tighe J, Laurent SJ, Bryant RA, Harvey SB. Road to resilience: a systematic review and meta-analysis of resilience training programmes and interventions. BMJ Open. 2018 Jun 14;8(6):e017858. doi: 10.1136/bmjopen-2017-017858. PMID 29903782
- [Background] Yehuda R, Flory JD, Southwick S, Charney DS. Developing an agenda for translational studies of resilience and vulnerability following trauma exposure. Ann N Y Acad Sci. 2006 Jul;1071:379-96. doi: 10.1196/annals.1364.028. PMID 16891584
- [Background] Palacio G C, Krikorian A, Gomez-Romero MJ, Limonero JT. Resilience in Caregivers: A Systematic Review. Am J Hosp Palliat Care. 2020 Aug;37(8):648-658. doi: 10.1177/1049909119893977. Epub 2019 Dec 13. PMID 31830813
- [Background] Terrill AL, Reblin M, MacKenzie JJ, Cardell B, Einerson J, Berg CA, Majersik JJ, Richards L. Development of a novel positive psychology-based intervention for couples post-stroke. Rehabil Psychol. 2018 Feb;63(1):43-54. doi: 10.1037/rep0000181. PMID 29553781
- [Background] O'Toole MS, Zachariae R, Renna ME, Mennin DS, Applebaum A. Cognitive behavioral therapies for informal caregivers of patients with cancer and cancer survivors: a systematic review and meta-analysis. Psychooncology. 2017 Apr;26(4):428-437. doi: 10.1002/pon.4144. Epub 2016 May 5. PMID 27147198
- [Background] Muller R, Gertz KJ, Molton IR, Terrill AL, Bombardier CH, Ehde DM, Jensen MP. Effects of a Tailored Positive Psychology Intervention on Well-Being and Pain in Individuals With Chronic Pain and a Physical Disability: A Feasibility Trial. Clin J Pain. 2016 Jan;32(1):32-44. doi: 10.1097/AJP.0000000000000225. PMID 25724020
- [Background] Casellas-Grau A, Font A, Vives J. Positive psychology interventions in breast cancer. A systematic review. Psychooncology. 2014 Jan;23(1):9-19. doi: 10.1002/pon.3353. Epub 2013 Jul 29. PMID 23897834
- [Background] Hausmann LR, Parks A, Youk AO, Kwoh CK. Reduction of bodily pain in response to an online positive activities intervention. J Pain. 2014 May;15(5):560-7. doi: 10.1016/j.jpain.2014.02.004. Epub 2014 Feb 22. PMID 24568751
- [Background] Cohn MA, Pietrucha ME, Saslow LR, Hult JR, Moskowitz JT. An online positive affect skills intervention reduces depression in adults with type 2 diabetes. J Posit Psychol. 2014 Jan 1;9(6):523-534. doi: 10.1080/17439760.2014.920410. PMID 25214877
- [Background] Moskowitz JT, Hult JR, Duncan LG, Cohn MA, Maurer S, Bussolari C, Acree M. A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test. J Health Psychol. 2012 Jul;17(5):676-92. doi: 10.1177/1359105311425275. Epub 2011 Oct 21. PMID 22021272
- [Background] Huffman JC, Mastromauro CA, Boehm JK, Seabrook R, Fricchione GL, Denninger JW, Lyubomirsky S. Development of a positive psychology intervention for patients with acute cardiovascular disease. Heart Int. 2011 Oct 3;6(2):e14. doi: 10.4081/hi.2011.e14. Print 2011 Sep 29. PMID 23825741
- [Background] Davidson F, Snow S, Hayden JA, Chorney J. Psychological interventions in managing postoperative pain in children: a systematic review. Pain. 2016 Sep;157(9):1872-1886. doi: 10.1097/j.pain.0000000000000636. PMID 27355184
- [Background] Charette S, Fiola JL, Charest MC, Villeneuve E, Theroux J, Joncas J, Parent S, Le May S. Guided Imagery for Adolescent Post-spinal Fusion Pain Management: A Pilot Study. Pain Manag Nurs. 2015 Jun;16(3):211-20. doi: 10.1016/j.pmn.2014.06.004. Epub 2014 Nov 6. PMID 25439116
- [Background] LaMontagne LL, Hepworth JT, Cohen F, Salisbury MH. Cognitive-behavioral intervention effects on adolescents' anxiety and pain following spinal fusion surgery. Nurs Res. 2003 May-Jun;52(3):183-90. doi: 10.1097/00006199-200305000-00008. PMID 12792259
- [Background] LaMontagne LL, Hepworth JT, Cohen F, Salisbury MH. Adolescent scoliosis: effects of corrective surgery, cognitive-behavioral interventions, and age on activity outcomes. Appl Nurs Res. 2004 Aug;17(3):168-77. doi: 10.1016/j.apnr.2004.06.007. PMID 15343550
- [Background] Richard HM, Nguyen DC, Podeszwa DA, De La Rocha A, Sucato DJ. Perioperative Interdisciplinary Intervention Contributes to Improved Outcomes of Adolescents Treated With Hip Preservation Surgery. J Pediatr Orthop. 2018 May/Jun;38(5):254-259. doi: 10.1097/BPO.0000000000000816. PMID 27328119
- [Background] Palermo TM, Lalloo C, Zhou C, Dampier C, Zempsky W, Badawy SM, Bakshi N, Ko YJ, Nishat F, Stinson JN. A cognitive-behavioral digital health intervention for sickle cell disease pain in adolescents: a randomized, controlled, multicenter trial. Pain. 2024 Jan 1;165(1):164-176. doi: 10.1097/j.pain.0000000000003009. Epub 2023 Sep 21. PMID 37733479
- [Background] Szeverenyi C, Kekecs Z, Johnson A, Elkins G, Csernatony Z, Varga K. The Use of Adjunct Psychosocial Interventions Can Decrease Postoperative Pain and Improve the Quality of Clinical Care in Orthopedic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Pain. 2018 Nov;19(11):1231-1252. doi: 10.1016/j.jpain.2018.05.006. Epub 2018 May 25. PMID 29803669
- [Background] Hohenschurz-Schmidt D, Vase L, Scott W, Annoni M, Ajayi OK, Barth J, Bennell K, Berna C, Bialosky J, Braithwaite F, Finnerup NB, Williams ACC, Carlino E, Cerritelli F, Chaibi A, Cherkin D, Colloca L, Cote P, Darnall BD, Evans R, Fabre L, Faria V, French S, Gerger H, Hauser W, Hinman RS, Ho D, Janssens T, Jensen K, Johnston C, Juhl Lunde S, Keefe F, Kerns RD, Koechlin H, Kongsted A, Michener LA, Moerman DE, Musial F, Newell D, Nicholas M, Palermo TM, Palermo S, Peerdeman KJ, Pogatzki-Zahn EM, Puhl AA, Roberts L, Rossettini G, Tomczak Matthiesen S, Underwood M, Vaucher P, Vollert J, Wartolowska K, Weimer K, Werner CP, Rice ASC, Draper-Rodi J. Recommendations for the development, implementation, and reporting of control interventions in efficacy and mechanistic trials of physical, psychological, and self-management therapies: the CoPPS Statement. BMJ. 2023 May 25;381:e072108. doi: 10.1136/bmj-2022-072108. No abstract available. PMID 37230508
- [Background] Zhou T, Luo Y, Xiong W, Meng Z, Zhang H, Zhang J. Problem-Solving Skills Training for Parents of Children With Chronic Health Conditions: A Systematic Review and Meta-Analysis. JAMA Pediatr. 2024 Mar 1;178(3):226-236. doi: 10.1001/jamapediatrics.2023.5753. PMID 38165710
- [Background] Basch E, Schrag D, Henson S, Jansen J, Ginos B, Stover AM, Carr P, Spears PA, Jonsson M, Deal AM, Bennett AV, Thanarajasingam G, Rogak LJ, Reeve BB, Snyder C, Bruner D, Cella D, Kottschade LA, Perlmutter J, Geoghegan C, Samuel-Ryals CA, Given B, Mazza GL, Miller R, Strasser JF, Zylla DM, Weiss A, Blinder VS, Dueck AC. Effect of Electronic Symptom Monitoring on Patient-Reported Outcomes Among Patients With Metastatic Cancer: A Randomized Clinical Trial. JAMA. 2022 Jun 28;327(24):2413-2422. doi: 10.1001/jama.2022.9265. PMID 35661856
- [Background] Jaensson M, Dahlberg K, Eriksson M, Nilsson U. Evaluation of postoperative recovery in day surgery patients using a mobile phone application: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1030-1038. doi: 10.1093/bja/aex331. PMID 29077818
- [Background] Sun X, Haydel KF, Matheson D, Desai M, Robinson TN. Are mobile phone ownership and age of acquisition associated with child adjustment? A 5-year prospective study among low-income Latinx children. Child Dev. 2023 Jan;94(1):303-314. doi: 10.1111/cdev.13851. Epub 2022 Sep 2. PMID 36056573
- [Background] Young NL, Varni JW, Snider L, McCormick A, Sawatzky B, Scott M, King G, Hetherington R, Sears E, Nicholas D. The Internet is valid and reliable for child-report: an example using the Activities Scale for Kids (ASK) and the Pediatric Quality of Life Inventory (PedsQL). J Clin Epidemiol. 2009 Mar;62(3):314-20. doi: 10.1016/j.jclinepi.2008.06.011. Epub 2008 Oct 1. PMID 18834710
- [Background] Moreno MA. Your Child's First Cell Phone. JAMA Pediatr. 2017 Jun 1;171(6):608. doi: 10.1001/jamapediatrics.2016.3115. No abstract available. PMID 28586792
- [Background] Brown SES, Costa C, Kelly A, et al. Adolescent and Caregiver Recovery Experiences After Minor Outpatient Surgery. Presented at: International Anesthesiology Research Society; May 2024; Seattle, WA.
- [Background] Woods SB, Roberson PNE, Booker Q, Wood BL, Booker SQ. Longitudinal Associations of Family Relationship Quality With Chronic Pain Incidence and Persistence Among Aging African Americans. J Gerontol B Psychol Sci Soc Sci. 2024 Jul 1;79(7):gbae064. doi: 10.1093/geronb/gbae064. PMID 38767217
- [Background] Psihogios AM, Schwartz LA, Ewing KB, Czerniecki B, Kersun LS, Pai ALH, Deatrick JA, Barakat LP. Adherence to Multiple Treatment Recommendations in Adolescents and Young Adults with Cancer: A Mixed Methods, Multi-Informant Investigation. J Adolesc Young Adult Oncol. 2020 Dec;9(6):651-661. doi: 10.1089/jayao.2020.0013. Epub 2020 May 11. PMID 32392434
- [Background] Psihogios AM, Fellmeth H, Schwartz LA, Barakat LP. Family Functioning and Medical Adherence Across Children and Adolescents With Chronic Health Conditions: A Meta-Analysis. J Pediatr Psychol. 2019 Jan 1;44(1):84-97. doi: 10.1093/jpepsy/jsy044. PMID 29982694
- [Background] Brown SES, Costa C, Kelly A, Oh S, Waitzman G, Dinh D, Clauw D, Waljee JF, Carlozzi NE. A Qualitative Assessment of Adolescent Symptom Report and Caregiver Concordance Following Outpatient Surgery. Clin J Pain. 2025 Jan 1;41(1):e1255. doi: 10.1097/AJP.0000000000001255. PMID 39668787
- [Background] Lima LACN, Otis A, Balram S, Giasson AB, Carnevale FA, Frigon C, Brown KA. Parents' perspective on recovery at home following adenotonsillectomy: a prospective single-centre qualitative analysis. Can J Anaesth. 2023 Jul;70(7):1202-1215. doi: 10.1007/s12630-023-02479-2. Epub 2023 May 9. PMID 37160822
- [Background] Cagiran E, Sergin D, Deniz MN, Tanatti B, Emiroglu N, Alper I. Effects of sociodemographic factors and maternal anxiety on preoperative anxiety in children. J Int Med Res. 2014 Apr;42(2):572-80. doi: 10.1177/0300060513503758. Epub 2014 Feb 5. PMID 24501165
- [Background] McGraw T. Preparing children for the operating room: psychological issues. Can J Anaesth. 1994 Nov;41(11):1094-103. doi: 10.1007/BF03015661. PMID 7828259
- [Background] Caumo W, Broenstrub JC, Fialho L, Petry SM, Brathwait O, Bandeira D, Loguercio A, Ferreira MB. Risk factors for postoperative anxiety in children. Acta Anaesthesiol Scand. 2000 Aug;44(7):782-9. doi: 10.1034/j.1399-6576.2000.440703.x. PMID 10939690
- [Background] Stanzel A, Sierau S. Pediatric Medical Traumatic Stress (PMTS) following Surgery in Childhood and Adolescence: a Systematic Review. J Child Adolesc Trauma. 2021 Aug 21;15(3):795-809. doi: 10.1007/s40653-021-00391-9. eCollection 2022 Sep. PMID 35958723
- [Background] Stargatt R, Davidson AJ, Huang GH, Czarnecki C, Gibson MA, Stewart SA, Jamsen K. A cohort study of the incidence and risk factors for negative behavior changes in children after general anesthesia. Paediatr Anaesth. 2006 Aug;16(8):846-59. doi: 10.1111/j.1460-9592.2006.01869.x. PMID 16884468
- [Background] Kotiniemi LH, Ryhanen PT, Moilanen IK. Behavioural changes in children following day-case surgery: a 4-week follow-up of 551 children. Anaesthesia. 1997 Oct;52(10):970-6. doi: 10.1111/j.1365-2044.1997.202-az0337.x. PMID 9370839
- [Background] Kaul P, Fisher MM. Addressing Key Issues in Adolescent Health Care. Pediatrics. 2020 May;145(Suppl 2):S151-S152. doi: 10.1542/peds.2019-2056B. No abstract available. PMID 32358205
- [Background] Kazak AE, Alderfer M, Rourke MT, Simms S, Streisand R, Grossman JR. Posttraumatic stress disorder (PTSD) and posttraumatic stress symptoms (PTSS) in families of adolescent childhood cancer survivors. J Pediatr Psychol. 2004 Apr-May;29(3):211-9. doi: 10.1093/jpepsy/jsh022. PMID 15131138
- [Background] Roth-Isigkeit A, Thyen U, Stoven H, Schwarzenberger J, Schmucker P. Pain among children and adolescents: restrictions in daily living and triggering factors. Pediatrics. 2005 Feb;115(2):e152-62. doi: 10.1542/peds.2004-0682. PMID 15687423
- [Background] Rosenbloom BN, Rabbitts JA, Palermo TM. A developmental perspective on the impact of chronic pain in late adolescence and early adulthood: implications for assessment and intervention. Pain. 2017 Sep;158(9):1629-1632. doi: 10.1097/j.pain.0000000000000888. No abstract available. PMID 28267063
- [Background] Palermo TM, de la Vega R, Murray C, Law E, Zhou C. A digital health psychological intervention (WebMAP Mobile) for children and adolescents with chronic pain: results of a hybrid effectiveness-implementation stepped-wedge cluster randomized trial. Pain. 2020 Dec;161(12):2763-2774. doi: 10.1097/j.pain.0000000000001994. PMID 32658147
- [Background] Fortier MA, Bunzli E, Walthall J, Olshansky E, Saadat H, Santistevan R, Mayes L, Kain ZN. Web-based tailored intervention for preparation of parents and children for outpatient surgery (WebTIPS): formative evaluation and randomized controlled trial. Anesth Analg. 2015 Apr;120(4):915-22. doi: 10.1213/ANE.0000000000000632. PMID 25790213
- [Background] Murray CB, Bartlett A, Meyyappan A, Palermo TM, Aaron R, Rabbitts J. A pilot feasibility and acceptability study of an Internet-delivered psychosocial intervention to reduce postoperative pain in adolescents undergoing spinal fusion. Can J Pain. 2022 Apr 13;6(1):12-23. doi: 10.1080/24740527.2021.2009334. eCollection 2022. PMID 35434455
- [Background] Gornitzky A, O'Donnell J, Diab M. More Than Just Medication: Exploring the Potential of a Perioperative Psychosocial Intervention Following Major Pediatric Orthopaedic Surgery. J Pediatr Soc North Am. 2024 Feb 12;5(2):592. doi: 10.55275/JPOSNA-2023-592. eCollection 2023 May. PMID 40433518
- [Background] Dussel V, Orellana L, Soto N, Chen K, Ullrich C, Kang TI, Geyer JR, Feudtner C, Wolfe J. Feasibility of Conducting a Palliative Care Randomized Controlled Trial in Children With Advanced Cancer: Assessment of the PediQUEST Study. J Pain Symptom Manage. 2015 Jun;49(6):1059-69. doi: 10.1016/j.jpainsymman.2014.12.010. Epub 2015 Jan 30. PMID 25640275
- [Background] Wolfe J, Orellana L, Cook EF, Ullrich C, Kang T, Geyer JR, Feudtner C, Weeks JC, Dussel V. Improving the care of children with advanced cancer by using an electronic patient-reported feedback intervention: results from the PediQUEST randomized controlled trial. J Clin Oncol. 2014 Apr 10;32(11):1119-26. doi: 10.1200/JCO.2013.51.5981. Epub 2014 Mar 10. PMID 24616307
- [Background] Palermo TM, Zempsky WT, Dampier CD, Lalloo C, Hundert AS, Murphy LK, Bakshi N, Stinson JN. iCanCope with Sickle Cell Pain: Design of a randomized controlled trial of a smartphone and web-based pain self-management program for youth with sickle cell disease. Contemp Clin Trials. 2018 Nov;74:88-96. doi: 10.1016/j.cct.2018.10.006. Epub 2018 Oct 11. PMID 30316999
- [Background] Lau N, Waldbaum S, Parigoris R, O'Daffer A, Walsh C, Colt SF, Yi-Frazier JP, Palermo TM, McCauley E, Rosenberg AR. eHealth and mHealth Psychosocial Interventions for Youths With Chronic Illnesses: Systematic Review. JMIR Pediatr Parent. 2020 Nov 10;3(2):e22329. doi: 10.2196/22329. PMID 33075743
- [Background] Rhodes L, Nash C, Moisan A, Scott DC, Barkoh K, Warner WC Jr, Sawyer JR, Kelly DM. Does preoperative orientation and education alleviate anxiety in posterior spinal fusion patients? A prospective, randomized study. J Pediatr Orthop. 2015 Apr-May;35(3):276-9. doi: 10.1097/BPO.0000000000000260. PMID 25036417
- [Background] LaMontagne L, Hepworth JT, Salisbury MH, Cohen F. Effects of coping instruction in reducing young adolescents' pain after major spinal surgery. Orthop Nurs. 2003 Nov-Dec;22(6):398-403. doi: 10.1097/00006416-200311000-00005. PMID 14705469
- [Background] Aust H, Eberhart L, Sturm T, Schuster M, Nestoriuc Y, Brehm F, Rusch D. A cross-sectional study on preoperative anxiety in adults. J Psychosom Res. 2018 Aug;111:133-139. doi: 10.1016/j.jpsychores.2018.05.012. Epub 2018 May 22. PMID 29935747
- [Background] Guite JW, McCue RL, Sherker JL, Sherry DD, Rose JB. Relationships among pain, protective parental responses, and disability for adolescents with chronic musculoskeletal pain: the mediating role of pain catastrophizing. Clin J Pain. 2011 Nov-Dec;27(9):775-81. doi: 10.1097/AJP.0b013e31821d8fb4. PMID 21593664
- [Background] Page MG, Campbell F, Isaac L, Stinson J, Katz J. Parental risk factors for the development of pediatric acute and chronic postsurgical pain: a longitudinal study. J Pain Res. 2013 Sep 30;6:727-41. doi: 10.2147/JPR.S51055. eCollection 2013. PMID 24109194
- [Background] Caes L, Vervoort T, Devos P, Verlooy J, Benoit Y, Goubert L. Parental distress and catastrophic thoughts about child pain: implications for parental protective behavior in the context of child leukemia-related medical procedures. Clin J Pain. 2014 Sep;30(9):787-99. doi: 10.1097/AJP.0000000000000028. PMID 24042348
- [Background] Birnie KA, Chorney J, El-Hawary R; PORSCHE Study Group. Child and parent pain catastrophizing and pain from presurgery to 6 weeks postsurgery: examination of cross-sectional and longitudinal actor-partner effects. Pain. 2017 Oct;158(10):1886-1892. doi: 10.1097/j.pain.0000000000000976. PMID 28598902
- [Background] Knoetze R, Lachman A, Moxley K, Chetty S. Caregiver anxiety and the association with acute postoperative pain in children undergoing elective ambulatory surgery in a lower-middle-income country setting. Paediatr Anaesth. 2020 Sep;30(9):990-997. doi: 10.1111/pan.13954. Epub 2020 Jul 9. PMID 32592506
- [Background] Vig A, Rathod KJ, Goel A, Nayak S, Jadhav AS, Pathak M, Saxena R, Sinha A. The understated issue of caregiver anxiety for pediatric surgical hospital admissions: opening the blindfolds. Pediatr Surg Int. 2023 Feb 3;39(1):100. doi: 10.1007/s00383-023-05380-7. PMID 36735080
- [Background] Rabbitts JA, Kain Z. Perioperative Care for Adolescents Undergoing Major Surgery: A Biopsychosocial Conceptual Framework. Anesth Analg. 2019 Oct;129(4):1181-1184. doi: 10.1213/ANE.0000000000004048. No abstract available. PMID 30720491
- [Background] Chow ET, Otis JD, Simons LE. The Longitudinal Impact of Parent Distress and Behavior on Functional Outcomes Among Youth With Chronic Pain. J Pain. 2016 Jun;17(6):729-38. doi: 10.1016/j.jpain.2016.02.014. Epub 2016 Mar 15. PMID 26993960
- [Background] Rabbitts JA, Fisher E. Postsurgical pain in children: unraveling the interplay between child and parent psychosocial factors. Pain. 2017 Oct;158(10):1847-1848. doi: 10.1097/j.pain.0000000000001000. No abstract available. PMID 28930920
- [Background] Caes L, Vervoort T, Eccleston C, Vandenhende M, Goubert L. Parental catastrophizing about child's pain and its relationship with activity restriction: the mediating role of parental distress. Pain. 2011 Jan;152(1):212-222. doi: 10.1016/j.pain.2010.10.037. Epub 2010 Dec 3. PMID 21126822
- [Background] Sarkisova N, Andras LM, Yang J, Tolo VT, Skaggs DL. High Parental Anxiety Increases Narcotic Use in Adolescent Patients Following Spinal Fusion. J Pediatr Orthop. 2020 Oct;40(9):e794-e797. doi: 10.1097/BPO.0000000000001549. PMID 32235191
- [Background] Rheel E, Ickmans K, Caes L, Vervoort T. The Impact of Parental Pain-attending and Non-pain-attending Responses on Child Pain Behavior in the Context of Cancer-related Painful Procedures: The Moderating Role of Parental Self-oriented Distress. Clin J Pain. 2021 Mar 1;37(3):177-185. doi: 10.1097/AJP.0000000000000902. PMID 33273274
- [Background] Eccleston C, Fisher EA, Vervoort T, Crombez G. Worry and catastrophizing about pain in youth: a reappraisal. Pain. 2012 Aug;153(8):1560-1562. doi: 10.1016/j.pain.2012.02.039. Epub 2012 Apr 18. No abstract available. PMID 22516589
- [Background] Page MG, Stinson J, Campbell F, Isaac L, Katz J. Pain-related psychological correlates of pediatric acute post-surgical pain. J Pain Res. 2012;5:547-58. doi: 10.2147/JPR.S36614. Epub 2012 Nov 12. PMID 23204864
- [Background] Rabbitts JA, Zhou C, Groenewald CB, Durkin L, Palermo TM. Trajectories of postsurgical pain in children: risk factors and impact of late pain recovery on long-term health outcomes after major surgery. Pain. 2015 Nov;156(11):2383-2389. doi: 10.1097/j.pain.0000000000000281. PMID 26381701
- [Background] Rabbitts JA, Palermo TM, Lang EA. A Conceptual Model of Biopsychosocial Mechanisms of Transition from Acute to Chronic Postsurgical Pain in Children and Adolescents. J Pain Res. 2020 Nov 24;13:3071-3080. doi: 10.2147/JPR.S239320. eCollection 2020. PMID 33262642
- [Background] Andersson V, Bergstrand J, Engstrom A, Gustafsson S. The Impact of Preoperative Patient Anxiety on Postoperative Anxiety and Quality of Recovery After Orthopaedic Surgery. J Perianesth Nurs. 2020 Jun;35(3):260-264. doi: 10.1016/j.jopan.2019.11.008. Epub 2020 Mar 5. PMID 32147278
- [Background] Theunissen M, Peters ML, Bruce J, Gramke HF, Marcus MA. Preoperative anxiety and catastrophizing: a systematic review and meta-analysis of the association with chronic postsurgical pain. Clin J Pain. 2012 Nov-Dec;28(9):819-41. doi: 10.1097/AJP.0b013e31824549d6. PMID 22760489
- [Background] Larach DB, Sahara MJ, As-Sanie S, Moser SE, Urquhart AG, Lin J, Hassett AL, Wakeford JA, Clauw DJ, Waljee JF, Brummett CM. Patient Factors Associated With Opioid Consumption in the Month Following Major Surgery. Ann Surg. 2021 Mar 1;273(3):507-515. doi: 10.1097/SLA.0000000000003509. PMID 31389832
- [Background] Yang MMH, Hartley RL, Leung AA, Ronksley PE, Jette N, Casha S, Riva-Cambrin J. Preoperative predictors of poor acute postoperative pain control: a systematic review and meta-analysis. BMJ Open. 2019 Apr 1;9(4):e025091. doi: 10.1136/bmjopen-2018-025091. PMID 30940757
- [Background] Nguyen SN, Hassett AL, Hu HM, Brummett CM, Bicket MC, Carlozzi NE, Waljee JF. Prospective cohort study on the trajectory and association of perioperative anxiety and postoperative opioid-related outcomes. Reg Anesth Pain Med. 2022 Oct;47(10):637-642. doi: 10.1136/rapm-2022-103742. Epub 2022 Aug 16. PMID 35973779
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Hassett AL, Hilliard PE, Goesling J, Clauw DJ, Harte SE, Brummett CM. Reports of chronic pain in childhood and adolescence among patients at a tertiary care pain clinic. J Pain. 2013 Nov;14(11):1390-7. doi: 10.1016/j.jpain.2013.06.010. Epub 2013 Sep 7. PMID 24021576
- [Background] Rabbitts JA, Fisher E, Rosenbloom BN, Palermo TM. Prevalence and Predictors of Chronic Postsurgical Pain in Children: A Systematic Review and Meta-Analysis. J Pain. 2017 Jun;18(6):605-614. doi: 10.1016/j.jpain.2017.03.007. Epub 2017 Mar 29. PMID 28363861
- [Background] Groenewald CB, Rabbitts JA, Schroeder DR, Harrison TE. Prevalence of moderate-severe pain in hospitalized children. Paediatr Anaesth. 2012 Jul;22(7):661-8. doi: 10.1111/j.1460-9592.2012.03807.x. Epub 2012 Feb 15. PMID 22332912
- [Background] Ellyson AM, Gordon G, Zhou C, Rabbitts JA. Trajectories, Risk Factors, and Impact of Persistent Pain After Major Musculoskeletal Surgery in Adolescents: A Replication Study. J Pain. 2022 Jun;23(6):995-1005. doi: 10.1016/j.jpain.2021.12.009. Epub 2021 Dec 31. PMID 34974171
- [Background] Rabbitts JA, Groenewald CB, Tai GG, Palermo TM. Presurgical psychosocial predictors of acute postsurgical pain and quality of life in children undergoing major surgery. J Pain. 2015 Mar;16(3):226-34. doi: 10.1016/j.jpain.2014.11.015. Epub 2014 Dec 22. PMID 25540939
- [Background] Tzong KY, Han S, Roh A, Ing C. Epidemiology of pediatric surgical admissions in US children: data from the HCUP kids inpatient database. J Neurosurg Anesthesiol. 2012 Oct;24(4):391-5. doi: 10.1097/ANA.0b013e31826a0345. PMID 23076227
- [Background] Rabbitts JA, Groenewald CB. Epidemiology of Pediatric Surgery in the United States. Paediatr Anaesth. 2020 Oct;30(10):1083-1090. doi: 10.1111/pan.13993. Epub 2020 Aug 29. PMID 32777147